CLINICAL TRIAL: NCT02471456
Title: Major Adverse Cardiac and Cerebrovascular Event (MACCE) & Patients' Quality of Life (QOL) After Endoscopic Vein Harvesting as Compared to Open Vein Harvest for Coronary Artery Bypass Grafting
Brief Title: MACCE After Endoscopic Vein Harvest for CABG
Acronym: MAQEH
Status: Completed | Type: Observational
Sponsor: The Royal Wolverhampton Hospitals NHS Trust (Other Government)
Collaborators: Maquet Cardiovascular (Industry)
Responsible Party: Sponsor
Other Study IDs: 2015CAR76
Record Dates: First submitted 2015-06-09; First posted 2015-06-15 (Estimated); Last update posted 2017-06-21 (Actual); Status verified 2017-06

CONDITIONS: Complications Due to Coronary Artery Bypass Graft

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- EVH: Patients that have undergone Endoscopic Vein Harvesting (EVH)
  Interventions: Other: Quality of Life Questionnaire; Other: MACCE review
- OVH: Patients that have undergone open vein harvest (OVH)
  Interventions: Other: Quality of Life Questionnaire; Other: MACCE review

INTERVENTIONS:
Other: Quality of Life Questionnaire — Quality of Life Questionnaire will be completed at least 1 year after their surgery.
Other: MACCE review — MACCE will be assessed by contacting the patient's GP and/or Cardiologist at least 1 year after their surgery.

SUMMARY:
Most patients undergoing coronary artery bypass grafting (CABG) will require long saphenous vein (LSV) harvesting from the leg. This has been reported to be associated with a significant morbidity (leg swelling, pain, infection, bruising, wound discharge) in up to 50% of patients. Endoscopic vein harvesting (EVH) which has been reported to be associated with a reduction in these complications was implemented within the investigators' service in 2012. Although some initial reports of concerns regarding graft patency when the LSV is harvested by EVH, NICE and European Cardiology Society (ESC/EACTS) guidelines 2014 supported the use of the EVH technology. Last year a service evaluation in the investigators' department showed significant cost benefit of EVH as compared to open vein harvest (OVH) in a matched group (50 EVH and 50 OVH patients). The purpose of this study is to evaluate this group further to assess the incidence of MACCE (Major adverse cardiac and cerebrovascular event) and patient's quality of life (QOL) at least 1 year after their surgery. MACCE will be assessed by contacting the patient's GP and/or Cardiologist and QOL questionnaire (SF12v2) will be sent to patients along with a patient information sheet. It is estimated that data collection would be completed within 3 months of start.

ELIGIBILITY:
Inclusion Criteria:

1. Patient underwent CABG (isolated or combined) during period Jan 2012 to Dec 2013
2. LSV harvested by EVH (Study group)
3. LSV Harvested by OVH matched with EVH group (Control group)

Exclusion Criteria:

1. Patient deceased at time of study start

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Fifty patients who underwent EVH (Study group) were part of our service evaluation when EVH was introduced to our practice. These patients were matched with patients undergoing CABG during the same period but where the LSV was harvested by OVH (50 patients, control group).
  This service evaluation showed a significant cost benefit when EVH was used in terms of reduction in the inhopsital stay, leg wound pain, leg wound infection and need to attend wound clinic. The current study is an extension of the service evaluation to assess how these patients are doing at least a year after their surgery in terms of MACCE, QOL,return to normal activities and survival
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2015-10-16 (Actual); Study Completion 2015-10-16 (Actual)

PRIMARY OUTCOMES:
MACCE in patients undergoing CABG where the LSV is harvested by EVH as compared to OVH | approximately 1 year
  The review of MACCE will occur at least 1 year after the patient's operation

SECONDARY OUTCOMES:
QOL as assessed by the SF12v2 questionnaire | approximately 1 year
  The review of QOL will occur at least 1 year after the patient's operation
Time taken to return to regular daily activities | approximately 1 year
  The review of time taken to return to regular daily activities will occur at least 1 year after the patient's operation
Survival | at approximately 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Heyman Luckraz, Principal Investigator — The Royal Wolverhampton NHS Trust
Locations (1):
- The Royal Wolverhampton NHS Trust, Wolverhampton, United Kingdom